CLINICAL TRIAL: NCT04281290
Title: Electrochemotherapy of Posterior Resection Surface for Lowering Disease Recurrence Rate in Pancreatic Cancer
Brief Title: Electrochemotherapy of Posterior Resection Surface for Lowering Disease Recurrence Rate in Pancreatic Cancer (PanECT Study)
Acronym: PanECT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After enrolling 3 participants the safety and efficacy of the planned treatment is questionable, thus we decided to terminate the study.
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Institute of Oncology Ljubljana (Other)
Responsible Party: Principal Investigator, Masa Bosnjak, Masa Bosnjak, PhD, researcher at Institute of Oncology Ljubljana (Collaborator), University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21K/01/20
Record Dates: First submitted 2020-01-14; First posted 2020-02-24 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pancreas Cancer
Keywords: Pancreatic cancer; Electrochemotherapy; Bleomycin
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Cliniporator Vitae® and chemotherapy drug Bleomycin PHC 15 e. (United States Pharmacopeia - USP)
  Interventions: Procedure: Electrochemotherapy - electroporation with Cliniporator Vitae® and chemotherapy drug Bleomycin PHC 15 e. (United States Pharmacopeia - USP)

INTERVENTIONS:
Procedure: Electrochemotherapy - electroporation with Cliniporator Vitae® and chemotherapy drug Bleomycin PHC 15 e. (United States Pharmacopeia - USP) — Procedure: Electrochemotherapy Exploration, anesthesia, pancreatic cancer resection, bleomycin administration, electroporation, formation of all anastomoses.
  Device: Cliniporator Vitae® Positioning of plate electrodes according to landmarks, 8-28 min after administration of bleomycin application of electric pulses (8 pulses, duration 100 microseconds, frequency 8 Hz with amplitude adequate to cover the whole treated lesion with electric field necessary for reversible plasma membrane permeabilization, approximately 1000V/cm), removal of electrodes.
  The maximum duration of procedure is 90 minutes, after liver mobilization.
  Drug: Bleomycin PHC 15 e. (United States Pharmacopeia - USP) Intravenous bolus administration of bleomycin (15 mg/m2)

SUMMARY:
The aim of the study is to evaluate toxicity and effectiveness of electrochemotherapy (ECT) with bleomycin in pancreatic cancer in clinical study phase I and II. After surgical resection of pancreatic cancer, the posterior resection surface will be treated with ECT with the intention to lower disease recurrence rate.

The study will include 20 patients in phase I clinical study and additional 20 patients in phase II clinical study (or in the extension of the clinical study), which will fulfill inclusion criteria.

Treatment effectiveness will be evaluated by US or CT imaging, to detect early local recurrence of the disease. Long term effectiveness of the treatment will be evaluated by frequent and precise patient follow-up. During follow-up clinical examination, laboratory tests, tumor markers (Ca 19-9 and CEA) and US/CT imaging will be performed.

The secondary objectives of the trial are to quantify the impact of the treatment on the patient's quality of life, tolerance to the therapy and suitability for larger study to be conducted.

DETAILED DESCRIPTION:
The study will be conducted on patients with resectable pancreatic cancer. 20 patients will be included in phase I clinical study and additional 20 patients in phase II clinical study (or in the extension of the clinical study).

After surgical resection of pancreatic cancer, the posterior resection surface will be treated with purpose to lower disease recurrence rate. Plate electrodes will be used for ECT treatment, the electrodes will be placed between choledochal cut-end, truncus celiacus, remaining of the pancreas and aortal lymph nodes.

ECT will be performed within 8-28 min after intravenous in bolus administration of bleomycin (15 mg/m2). Triggering of electric pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart.

All patients will be treated after the procedure has been thoroughly described to them and have signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable pancreatic cancer.
2. Histologically confirmed and/or based on radiological imaging and laboratory tests confirmed pancreatic cancer by multidisciplinary team for pancreatic tumors.
3. Age more than 18.
4. Life expectancy more than 3 months.
5. Performance status - Karnofsky ≥ 70 or WHO < or 2.
6. Treatment free interval 2-5 weeks, depending on the drugs used.
7. Patient must be mentally capable of understanding the information given.
8. Patient must give informed consent.
9. Patient must be discussed at the multidisciplinary team for pancreatic tumors before entering the trial.

Exclusion Criteria:

1. Secondary primary tumor, except surgically treated noninvasive cancer of cervix, or surgically or irradiated basal cell carcinoma.
2. Proven visceral, bone or diffuse metastases.
3. Life-threatening infection and/or heart failure and/or liver failure and/or renal failure (creatinine more than 150 µmol/L) other severe systemic pathologies.
4. Significant reduction in respiratory function.
5. Age less than 18 years.
6. Cumulative dose of 250 mg/m2 bleomycin received.
7. Allergic reaction to bleomycin.
8. Patients with epilepsy.
9. Patients with arrhythmias.
10. Patients with heart failure or pacemaker.
11. Pregnancy.
12. Patient incapable of understanding the aim of the study or disagree with the entering into the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of feasibility and safety | 7 days after operation
  Every patient will be closely followed-up after operation with clinical examination and blood tests (hemogram, comprehensive metabolic panel, liver panel) according to the study protocol (day 1, 3, 7 after operation). In case of detected abnormalities additional imaging (US and/or CT) will take place. Findings will be noted and reported in line with Clavien-Dindo classification of surgical complications. The primary measure is to detect complications after surgery and to determine whether the complication is related to electrochemotherapy treatment or not.

SECONDARY OUTCOMES:
Disease-free Survival | 1, 3, 6, 12, 18 and 24 months after operation
  Disease-free survival is defined as the amount of time a subject survives without disease recurrence after treatment. Recurrence is defined as significant elevation of tumor markers Ca19-9 and CEA after operation (normal value of Ca19-9 is under 37.0 kU/L, normal value of CEA is under 4.2 µg/L). The appearance of one or more lesions on imaging investigation (US and/or CT) is also considered a recurrence.
  The tumor markers and imaging investigations will be performed according to study protocol (tumor markers 1, 3, 6, 12 and 24 months after operation; imaging 1, 3, 6, 12, 18 and 24 months after operation - the imaging method will be CT or MR with or without contrast, with the exception of 1 and 18 months after the operation when an US will be performed).
Overall Survival | From the time of surgical treatment until 5 years after surgery
  Overall survival is defined as the amount of time a subject survives after therapy. Patient enrolled in the study will be followed up for at least five years. During first two years after surgery follow-up will be as written above, after that period patient will be followed-up according every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mihajlo Djokic, MD, PhD, Principal Investigator — University Medical Centre Ljubljana, Ljubljana, Slovenia; Blaz Trotovsek, MD, PhD, Study Director — University Medical Centre Ljubljana, Ljubljana, Slovenia; Gregor Sersa, PhD, Study Director — Institute of Oncology, Ljubljana, Slovenia; Zan Cebron, MD, Study Chair — University Medical Centre Ljubljana, Ljubljana, Slovenia; Miha Petric, MD, Study Chair — University Medical Centre Ljubljana, Ljubljana, Slovenia; David Badovinac, MD, Study Chair — University Medical Centre Ljubljana, Ljubljana, Slovenia; Masa Bosnjak, PhD, Study Chair — Institute of Oncology, Ljubljana, Slovenia; Bostjan Markelc, PhD, Study Chair — Institute of Oncology, Ljubljana, Slovenia; Maja Cemazar, PhD, Study Chair — Institute of Oncology, Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Djokic M, Cemazar M, Popovic P, Kos B, Dezman R, Bosnjak M, Zakelj MN, Miklavcic D, Potrc S, Stabuc B, Tomazic A, Sersa G, Trotovsek B. Electrochemotherapy as treatment option for hepatocellular carcinoma, a prospective pilot study. Eur J Surg Oncol. 2018 May;44(5):651-657. doi: 10.1016/j.ejso.2018.01.090. Epub 2018 Feb 2. PMID 29402556
- [Background] Bimonte S, Leongito M, Granata V, Barbieri A, Del Vecchio V, Falco M, Nasto A, Albino V, Piccirillo M, Palaia R, Amore A, Giacomo Rd, Lastoria S, Setola SV, Fusco R, Petrillo A, Izzo F. Electrochemotherapy in pancreatic adenocarcinoma treatment: pre-clinical and clinical studies. Radiol Oncol. 2016 Feb 16;50(1):14-20. doi: 10.1515/raon-2016-0003. eCollection 2016 Mar 1. PMID 27069445
- [Background] Tafuto S, von Arx C, De Divitiis C, Maura CT, Palaia R, Albino V, Fusco R, Membrini M, Petrillo A, Granata V, Izzo F; ENETS Center of Excellence Multidisciplinary Group for Neuroendocrine Tumors in Naples (Italy). Electrochemotherapy as a new approach on pancreatic cancer and on liver metastases. Int J Surg. 2015 Sep;21 Suppl 1:S78-82. doi: 10.1016/j.ijsu.2015.04.095. Epub 2015 Jun 27. PMID 26123385